CLINICAL TRIAL: NCT04688710
Title: Use of Audio Recordings of Self-Hypnosis and Meditation for Fatigue Management in Multiple Sclerosis
Acronym: AUDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Mark Jensen, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011189; RG-2001-36025 (Other: National Multiple Sclerosis Society)
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Hypnosis; Mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized, 3-group parallel design, 333-subject clinical trial to test the efficacy of Self-Hypnosis (HYP) and Mindfulness Meditation (MM) compared to Treatment as Usual (TAU) for individuals with multiple sclerosis and clinically significant fatigue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Hypnosis (HYP) (Active Comparator): Participants receive an instructional manual and instructional audio recording to explain the study treatment and how to use audio recordings. Participants then receive a set of audio recordings once per week for 4 weeks teaching Self-Hypnosis. Following the 4 weeks of training to use treatment recordings, you will have 6 months of access to the recordings. Participants may access the recordings to use when convenient and are encouraged to access recordings daily for practice.
  Interventions: Behavioral: Self-Hypnosis (HYP)
- Mindfulness Meditation (MM) (Active Comparator): Participants receive an instructional manual and instructional audio recording to explain the study treatment and how to use audio recordings. Participants then receive a set of audio recordings once per week for 4 weeks teaching Mindfulness Meditation. Following the 4 weeks of training to use treatment recordings, you will have 6 months of access to the recordings. Participants may access the recordings to use when convenient and are encouraged to access recordings daily for practice.
  Interventions: Behavioral: Mindfulness Meditation (MM)
- Treatment as Usual (TAU) (No Intervention): Participants will not receive treatment from the study during the treatment phase. Participants will continue to receive their normal care outside of the study for MS and fatigue. Participants will have the option to access either the Self-Hypnosis or Mindfulness Meditation treatment after all study assessments have been completed.

INTERVENTIONS:
Behavioral: Self-Hypnosis (HYP) — Self-Hypnosis (HYP) teaches skills people with MS can use to effectively self-manage symptoms related to fatigue. Recordings are designed to help participants learn new strategies for influencing fatigue and its effects on their lives. The Self-Hypnosis recordings will start with a relaxation hypnotic induction (e.g., "Notice how with each breath, you are feeling more and more relaxed …") followed by hypnotic suggestions (e.g., for experiencing more energy, improved sleep, more comfort or less pain, etc.). The goal of Self-Hypnosis is to change participant's experiences. To the extent that participants respond to the suggestions, participants would then get more control over their feelings of energy, sleep quality, and comfort levels.
  Arms: Self-Hypnosis (HYP)
Behavioral: Mindfulness Meditation (MM) — Mindfulness Meditation (MM) teaches skills people with MS can use to effectively self-manage symptoms related to fatigue. Recordings are designed to help participants learn about a new way to live with chronic fatigue and new ways to relate to how fatigue may influence their thoughts, feelings, and behavior. The mindfulness techniques train the mind to non-judgmentally observe experience (e.g., symptoms of fatigue or pain, etc.) on a moment-to-moment basis, with an attitude of acceptance. The goal of Mindfulness Meditation is not to alter experiences, but rather to change how someone responds to their experiences. With practice, automatic, kneejerk reactions to symptoms are replaced with mindful choices about how best to respond to symptoms. This will "lighten the load" of living with the symptoms, moving participants in the valued direction of their choosing.
  Arms: Mindfulness Meditation (MM)

SUMMARY:
The purpose of this study is to assess the effectiveness of two self-guided psychological treatments, Self-Hypnosis (HYP) and Mindfulness Meditation (MM) compared to Treatment as Usual (TAU) for people with multiple sclerosis (MS) and clinically significant fatigue.

DETAILED DESCRIPTION:
People with multiple sclerosis (MS) often have problems with fatigue that can interfere with other treatments. As many as 90% of individuals with MS experience persistent fatigue and 40% of individuals with MS describe fatigue as their most debilitating symptom. Fatigue in individuals with MS is also associated with greater distress and lower overall quality of life. Unfortunately, available treatments provide inadequate relief for most people. There remains an urgent need for additional treatment options for MS-related fatigue. The purpose of this study is to see if self-guided psychological treatments delivered through audio recordings can help decrease fatigue severity in people with MS.

This study will evaluate the efficacy of two promising and innovative psychological treatments, Mindfulness Meditation (MM) and Self-Hypnosis (HYP), for helping individuals with MS manage fatigue. Since these treatments are self-guided, findings will provide evidence for the efficacy of highly accessible treatments, ultimately resulting in treatment interventions that can be easily disseminated without the need for highly trained specialist clinicians.

Primary Aim: The primary aim of the proposed research is to evaluate the beneficial effects of two treatments (HYP and MM) for reducing MS-related fatigue, relative to Treatment as Usual (TAU).

Primary Hypothesis (stated under the alternative): Participants assigned to HYP and MM conditions will report significantly greater reductions in fatigue at post-treatment, the primary end point, than those assigned to the TAU condition.

The proposed research also has three secondary aims:

Secondary Aim 1: To investigate whether there are beneficial effects of the two active treatments, relative to TAU, on pre- to post-treatment changes in secondary quality of life outcomes (e.g., sleep quality, pain intensity).

Secondary Aim 2: To investigate whether there are longer-term benefits of the two active treatments, relative to each other and to TAU, on the primary and secondary outcomes, up to 6 months post-treatment.

Exploratory Aim 3: To investigate whether there is participant preference for either of the two active treatments, and investigate their relative effects on the study outcomes in an "open label" effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported diagnosis of MS.
2. Age 18 years old or older at the time of study enrollment.
3. Presenting with clinically meaningful fatigue (i.e., reporting daily fatigue ≥50% of the days in the past 6 months with an average severity in the past week of ≥ 20 on the PROMIS Fatigue short form [T-score, 56.4]).
4. Able to read, speak, and understand English.
5. Access to an internet-enabled device (desktop/laptop/tablet/smart phone) to allow access to the recordings and to complete the study measures via the internet.

Exclusion Criteria:

1. Psychiatric condition or symptoms that would interfere with participation, specifically (a) current active suicidal ideation with current intent to harm oneself, (b) current psychosis, or (c) current mania.
2. Currently receiving psychological treatment for fatigue more than once per month.
3. Has received mindfulness meditation or hypnosis training in the past and has practiced mindfulness meditation/hypnosis in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Severity | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in fatigue severity will be measured using the Modified Fatigue Impact Scale (MFIS). The 21-item MFIS was selected as the measure of choice for assessing fatigue in MS populations by the MS Council for Clinical Practice Guidelines. The MFIS is also listed as one of the NIH NINDS' common data elements for MS. With the MFIS, respondents indicate the frequency with which they experience each fatigue-related outcome (e.g., forgetful, weak muscles) on a 5-point Likert scale (0 = Never; 4 = Almost always). The items can be scored into three subscales (reflecting cognitive, physical, and psychosocial fatigue impact) or a total fatigue severity score.

SECONDARY OUTCOMES:
Change in Sleep Quality assessed via PROMIS Sleep Disturbance Short Form 4a, version 1.0 | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in sleep quality will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 4a, version 1.0. Responses from each item will be summed to form a total raw score ranging from 4-20. Higher scores indicate higher self-reported levels of sleep disturbance.
Change in Pain Interference | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in pain interference will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 4a, version 1.1. Responses from each item will be summed to form a total raw score ranging from 4-20. Higher scores indicate higher self-reported levels of pain interference.
Change in Pain Intensity and Fatigue (current) | Immediately before and after listening to treatment audio recordings
  Change in current pain intensity and fatigue will be measured using a 0-10 numeric rating scale immediately before and after listening to audio recordings.
Change in Pain Intensity (past week) | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in pain intensity in the past week will be measured using a 0-10 numeric rating scale.
Change in Depressive Symptoms | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in depressive symptoms will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 4a, version 1.0. Responses from each item will be summed to form a total raw score ranging from 4-20. Higher scores indicate higher self-reported levels of depressive symptoms.
Change in Anxiety | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in symptoms of anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 4a, version 1.0. Responses from each item will be summed to form a total raw score ranging from 4-20. Higher scores indicate higher self-reported levels of anxiety symptoms.
Change in Physical Function | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in physical function will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 4a, version 2.0. Responses from each item will be summed to form a total raw score ranging from 4-20. Higher scores indicate higher self-reported levels of physical functioning.
Treatment Preference | Baseline (prior to treatment)
  Participants' preferences for each of the three randomization groups will be measured at baseline (prior to treatment). Treatment preferences will be measured using a 0 (not at all interested) - 10 (extremely interested) numerical rating scale to gauge interest in each randomization group.
Device Use for Treatment | Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Type of device(s) used to access treatment recordings will be assessed by participant self-report.
Change in Global Impression of Change | Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Global impression of change will be measured by participant self-report. Participants will report, since the start of the study, how much they think their overall fatigue intensity, interference of fatigue in daily activities, and ability to manage fatigue has changed on a scale of 1 (very much improved) - 7 (very much worse).
Change in Global Assessment of Treatment Satisfaction | Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Global assessment of treatment satisfaction will be measured by participant self-report on a scale of 0 (very dissatisfied) - 4 (very satisfied).
Barriers and Facilitators to Treatment | Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Barriers and facilitators to participants engaging in treatment will be assessed by qualitative open-ended questions asking what made it harder or easier for participants to listen to recordings, as well as what participants liked most and least about listening to recordings.

OTHER OUTCOMES:
Medication and/or Cannabis Use | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Medication use will be assessed by asking participants to report whether or not they are using any opioids, antidepressants, anticonvulsants, sedative/hypnotic, or NSAID medications or cannabinoids or marijuana products within the past 7 days.
Frequency and Duration of Listening to Treatment Audio Recordings | Each time treatment recordings are accessed from Week 1 through Week 24
  Frequency and duration of listening to treatment recordings will be logged by the software participants will use to access recordings. Treatment
Change in Fatigue Catastrophizing | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in pain catastrophizing will be measured with items from the University of Washington (UW) Concerns about Pain (UW CAP-6-SF), adapted for fatigue symptoms. The UW CAP-6-SF, adapted for fatigue is scored by summing item responses for a total raw score from 6-30. Higher scores indicate a higher level of fatigue catastrophizing.
Pain Type | Baseline (prior to treatment)
  Pain type will be assessed using the painDETECT Pain Questionnaire to assess for the presence of neuropathic pain. The painDETECT is scored by summing responses to each item to create a total raw score between 0-38, where a score of 0-12 indicates neuropathic pain component is unlikely (<15%), a score of 13-18 indicates the result is ambiguous and a neuropathic pain component can be present, and a score of 19-38 indicates a neuropathic pain component is likely (>90%).
Change in Pain Catastrophizing | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in fatigue catastrophizing will be measured with items from the University of Washington (UW) Concerns about Pain (UW CAP-2-SF). The UW CAP-2-SF, is scored by summing item responses for a total raw score from 2-10. The total raw score will then be converted to a IRT (Item Response Theory)-based T-score. Higher T scores indicate a higher level of pain catastrophizing. Higher scores indicate a higher level of pain catastrophizing.
Change in Readiness to Engage in Pain Self-Management | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Readiness to engage in pain self-management will be measured using the items/scales from the Multidimensional Pain Readiness to Change Questionnaire, Version 2 (MPRCQ2), with additional items about meditation and self-hypnosis. The MPRCQ2 is scored by summing the responses for each scale (e.g, exercise, relaxation, pacing, etc.) or sub scale and dividing by the number of items to get the mean response. Higher scores in each scale or sub scale indicates higher levels of that domain in regards to pain management.
Change in Pain-Related Cognitive Processes | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in pain-related cognitive processes will be assessed using the pain openness scales from the Pain-Related Cognitive Processes Questionnaire (PCPQ). The pain openness scales are scored by adding up items in the scale and dividing by number of items to completed to find the mean response. Higher scores indicate higher levels of pain openness.
Change in Satisfaction with Life assessed via the Satisfaction with Life Scale (SWLS) | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in satisfaction with life will be assessed using the Satisfaction with Life Scale (SWLS). The SWLS is scored by summing the items to create a total raw score from 5-35. Higher scores indicate higher satisfaction with life.
Change in Mindfulness | Baseline (prior to treatment), Week 4 (post-treatment), Week 12 (3 month follow-up), Week 24 (6-month follow-up)
  Change in mindfulness will be assessed using the 15-item Five-Facet Mindfulness Questionnaire (FFMQ-15). The FFMQ-15 is scored by summing items to create a total raw score from 15-75 with higher scores indicating higher levels of mindfulness.
Outcome Expectancy | Baseline (prior to treatment)
  Outcome expectancy refers to assessing participants' expectations regarding how logical and effective they believe the treatment they are randomized to receive will be prior to engaging in treatment. Participants' expectations regarding their outcomes are measured on a scale of 0-10 with higher scores indicating higher expectations for treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- UW Medicine Multiple Sclerosis Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data used for each paper published from the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. Proposals should be directed to Dr. Mark Jensen (mjensen@uw.edu). To gain access, requestors will need to sign a data access agreement. Data will be provided via a HIPAA-compliant file sharing system.